CLINICAL TRIAL: NCT04636736
Title: Possible Changes in HIV Drug Resistance Pattern Due to Migration of People From the Eastern Europe to Poland
Brief Title: HIV Drug Resistance Pattern Due to Migration in Poland
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrzej Załęski, Principal Investigator, Medical University of Warsaw
Other Study IDs: HIVresistancePL
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; HIV-1-infection; Resistant Infection
Keywords: HIV-infection; AIDS; migration; cART; drug-resistance
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — HIV- RNA and standard analysis of drug-resistance pattern
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV POLISH (PL): HIV infected people with polish nationality, who most probably acquired infection in Poland
  Interventions: Diagnostic Test: HIV drug resistance testing
- HIV MIGRANTS (M): HIV infected people, originating from outside of Poland, where they were diagnosed with HIV infection
  Interventions: Diagnostic Test: HIV drug resistance testing

INTERVENTIONS:
Diagnostic Test: HIV drug resistance testing — HIV drug resistance testing in people newly diagnosed in HIV in Poland

SUMMARY:
According to the Polish governmental statistics migration of people from Ukraine to Poland is growing and only in year 2020 have come to Poland about a quarter of a million of Ukrainian migrants. As well, more than 40% of those diagnosed with HIV infection in the European Union (EU)/European Economic Area (EEA) in 2018 were also migrants, originating from countries with generalized HIV epidemics, such as Ukraine. Antiretroviral treatment should be started, based, among others, on epidemiological data and evidence of presence of drug resistance mutations in a the population.

DETAILED DESCRIPTION:
BACKGROUND:

According to the Polish governmental statistics during the year 2020 have come to Poland about 240 thousand of ukarinian migrants, and it is estimated that nowadays in Poland live and work about 1.2 million of people from Ukraine. In recent years substantial increases in diagnosis of HIV infected people have been reported in some countries, including Poland. At the same time 42% of those diagnosed in the EU/EEA in 2018 were migrants, defined as originating from outside of the country in which they were diagnosed. More than one-third (40%) of newly diagnosed cases due to heterosexual transmission were among migrants originating from countries with generalized HIV epidemics, such as Ukraine. Overall in the EU/ EEA, and even in some settings with decrease in newly diagnosed HIV infections in men having sex with others men (MSM), new HIV diagnoses in migrant MSM have not declined at the same rate as those who are not foreign-born. Antiretroviral treatment should be started immediately in all HIV-positive patients, regardless of origin, race, gender or sexual preferences. The choose of first-line antiretroviral regimen is based, among others, on epidemiological data and evidence of presence of drug resistance mutations in a the population.

AIM OF THE STUDY:

Due to changes in epidemiological pattern in newly diagnosed patients with HIV infection in Poland and increase in number of HIV positive patients from Ukraine we aimed to asses whether the presence of drug resistance mutations in the population of Ukrainian patients differs from the pattern of resistance of not foreign born patients with newly diagnosed HIV infection in Poland. The potential differences may have further implications on antiretroviral regimens in drug naive HIV positive patients.

MATERIAL AND METHODS:

We have designed observational, prospective study which will be performed in several clinical centers in Poland. As a part of the study we will collect epidemiological (age, gender, origin, migration data, sexual preferences) and clinical data (HIV viral load, CD4+ cells count, presence of AIDS-defining diseases, proposed combined antiretrovirat therapy (cART) regimen and the response to the treatment, Hepatitis B (HBV) and C (HCV) co-infections).

In all patients, before starting antiretroviral treatment, presence of drug resistance mutations of HIV will be assessed. The molecular diagnostics will cover mutations to the nucleotide and non-nucleotide reverse transcriptase inhibitors (NRTI and NNRTI), protease inhibitors (PI) and as well integrase inhibitors (InSTI).

Statistical evaluation will be performed in subgroups of migrants and in patients born in Poland. The distribution of continuous variables will be analysed by the Shapiro-Wilk test. The data will be expressed as the median and interquartile range (IQR). Quantitative data will be analysed using the Mann-Whitney U test or Kruskal-Wallis ANOVA when appropriate. Qualitative data will be compared using the χ² test or the Fisher exact test. A P value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* recent diagnosis with HIV infection (<6 months)
* no history of antiretrovirals intake (PrEP, PEP)
* age 18 years or olde

Exclusion Criteria:

- failure to meet any of the inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People diagnosed with HIV infection in Poland, originating from Poland and other countries
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in HIV drug resistance pattern | 2 years
  Differences between people originating from Poland and from Eastern Europe

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Wiercińska-Drapało, PhD, Study Chair — Department of Infectious Diseases,Tropical Diseases and Hepatology, Medical University of Warsaw
Locations (1):
- Department of Infectious Diseases, Tropical Diseases and Hepatology, Medical University of Warsaw, Warsaw, Mazowia, Poland

IPD SHARING:
Plan to Share IPD: No
there is no plan to share the data

REFERENCES:
- [Background] Wensing AM, Calvez V, Ceccherini-Silberstein F, Charpentier C, Gunthard HF, Paredes R, Shafer RW, Richman DD. 2019 update of the drug resistance mutations in HIV-1. Top Antivir Med. 2019 Sep;27(3):111-121. PMID 31634862
- [Background] Shafer RW, Rhee SY, Pillay D, Miller V, Sandstrom P, Schapiro JM, Kuritzkes DR, Bennett D. HIV-1 protease and reverse transcriptase mutations for drug resistance surveillance. AIDS. 2007 Jan 11;21(2):215-23. doi: 10.1097/QAD.0b013e328011e691. PMID 17197813
- [Derived] Zaleski A, Lembas A, Dyda T, Siwak E, Osinska J, Suchacz M, Stempkowska-Rejek J, Strycharz M, Orzechowska J, Wiercinska-Drapalo A. Changes in Primary HIV-1 Drug Resistance Due to War Migration from Eastern Europe. J Immigr Minor Health. 2024 Feb;26(1):15-22. doi: 10.1007/s10903-023-01559-1. Epub 2023 Nov 16. PMID 37973713
- See also: Hiv surveillance report — https://ecdc.europa.eu/sites/default/files/documents/hiv-surveillance-report-2019.pdf
- See also: Migration report in Poland — https://migracje.gov.pl
- See also: Migration report in Poland — https://obserwatorfinansowy.pl/tematyka/makroekonomia/trendy-gospodarcze/nowa-fala-migracji-obywateli-ukrainy-do-polski/
- See also: Hiv resistance pattern — http://cms.hivdb.org/prod/downloads/resistance-mutation-handout/resistance-mutation-handout.pdf
- See also: HIV/AIDS European guidelines on diagnostics and treatment — https://eacsociety.org/files/2019_guidelines-10.0_final.pdf